CLINICAL TRIAL: NCT04557774
Title: Cognitive Function of Alcoholic Liver Disease Patients
Brief Title: Cognitive Function of Alcoholic Compensated Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Suk, Proffesor, Chuncheon Sacred Heart Hospital
Other Study IDs: COG; YR (Other: Hallym university)
Record Dates: First submitted 2020-09-08; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Alcoholic Liver Disease
Keywords: Hepatic encephalopathy; Liver cirrhosis; Cognition; Alcohol; BMI
MeSH Terms: conditions — Liver Diseases, Alcoholic; Hepatic Encephalopathy; Liver Cirrhosis | interventions — Neuropsychological Tests; Laboratories; X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver cirrhosis group: All included patients were asymptomatic at the baseline with no evidence of neurological impairment. Patients with a history of moderate alcohol drinking plus hepatitis B/C virus infection, medication for sedation, MELD (Model for End-stage Liver Disease) score of more than 20, OHE, seizure, head trauma, stroke, dementia, Parkinson's disease, or any kind of focal neurologic deficits were excluded. Any patients who were suspected of alcohol induced direct neurologic damages such as Wernicke's encephalopathy, alcohol induced spinal cord disease, or alcohol induced peripheral nerve disease were excluded. After evaluating the data including the laboratory findings, image findings, endoscopic findings, and medical records of all these patients, as well as liver biopsy findings for some patients, we sub-classified these 88 patients into two groups: alcoholic LC and viral LC. Finally, 80 patients (viral: 37; alcohol: 43) with compensated LC were prospectively considered in this study.
  Interventions: Other: Cognitive function test

INTERVENTIONS:
Other: Cognitive function test — Laboratory and imaging test
  * Biochemical serum test: total bilirubin, alanine aminotransferase (ALT), haptoglobin, aspartate aminotransferase (AST), gamma glutamyltranspeptidase (GGT), alkaline phosphatase (ALP), albumin, blood urea nitrogen, creatinine, α-fetoprotein (AFP), prothrombin time, blood glucose, triglycerides, and total cholesterol.
  * Baseline evaluations: family and alcohol history, X-ray, electrocardiography, blood tests for electrolyte, liver function, and viral markers
  Neuropsychological test
  -Attention, Language, Visuospatial, Memory, Frontal/executive
  Other Names: Laboratory, imaging, neuropsychological tests

SUMMARY:
Differences in cognitive function between patients with viral and alcoholic compensated liver cirrhosis

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is one of the important complications of liver cirrhosis (LC). HE exhibits alterations in cognitive, psychomotor-intellectual, emotional, behavioral, or fine-motor functions. Approximately 22-74 % of patients with non-fulminant HE have MHE with a frequency proportional to the patient age and the severity of the liver disease. Patients with MHE exhibit disability in most functional behaviors such as social connection, alertness, emotional behavior, sleep, work, and leisure.

Alcohol consumption itself has a toxic effect on the brain. It has been documented that there is a neuronal loss in the cerebral cortex, hypothalamus, hippocampus, septal region, and cerebellum of an alcoholic brain.

The major causes of LC are hepatitis B/C viral infection and chronic alcohol consumption. The most widely accepted theory of HE pathogenesis is that toxic substances derived from the gut affect cerebral function after liver dysfunction or portosystemic shunting. This proposed pathogenetic mechanism could apply to viral compensated LC. However, it is difficult to explain the development of MHE in patients with alcoholic LC in this manner.

Therefore, patients with alcoholic LC may have different cognitive dysfunction as compared to patients with viral LC.

ELIGIBILITY:
Inclusion Criteria:

* Those who agreed to participate in this study and signed a written consent
* Those who have no evidence of neurological impairment

Exclusion Criteria:

* Those who have decompensated liver cirrhosis
* Those who have a high MELD score (≥20)
* Those who have OHE during admission
* Those who have parients' refusal

Ages: 22 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All of them are agree to provide it to investigation.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2013-03-01 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Liver function | 10 years
  Compare the liver enzyme level Serum biochemical parameters included total bilirubin(mg/dL), alanine aminotransferase(ALT(IU/L)), haptoglobin(mg/dL), aspartate aminotransferase (AST (IU/L)), gamma glutamyltranspeptidase (GGT(IU/L)), alkaline phosphatase (ALP(IU/L)), albumin(g/dL), blood urea nitrogen(mg/dL), creatinine(mg/dL), α-fetoprotein (AFP(ng/mL)), prothrombin time, blood glucose(mg/dL), triglycerides(mg/dL), and total cholesterol(mg/dL).
Cognitive function (Neuropsychological test) | 10 years
  Assessment to measure cognitive function using neuropsychological test
BMI | 10 years
  Compare the body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Ki Tae Suk, Principal Investigator — Hallym University Medical Center
Locations (1):
- Department of Internal Medicine, Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwondo, South Korea

IPD SHARING:
Plan to Share IPD: No